CLINICAL TRIAL: NCT04858191
Title: Utilizing Hyperpolarized 129Xe Magnetic Resonance Imaging in Children With Primary Ciliary Dyskinesia
Acronym: PCD MRI
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Principle investigator, The Hospital for Sick Children
Other Study IDs: 1000068639
Record Dates: First submitted 2021-03-25; First posted 2021-04-26 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Xenon MRI; Lung; Pulmonary Exacerbation
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric PCD: Pediatric participants with PCD

SUMMARY:
This study investigates the use of hyperpolarized 129Xe magnetic resonance imaging (MRI) in children with primary ciliary dyskinesia (PCD) in detecting ventilation defects. The investigators will establish the feasibility and reliability of this test and how it changes compared to other pulmonary function tests.

DETAILED DESCRIPTION:
Primary Ciliary Dyskinesia (PCD) is an autosomal recessive inherited disorder caused by defects in ciliary structure and/or function. Prevention or delaying disease progression requires medical therapies and routine lung function monitoring, with the goal of early initiation of medical therapies. Of course, this is contingent on recognizing early lung disease.

Current investigations for monitoring lung disease include pulmonary function tests (PFT), chest x rays and chest CTs. But each of these modalities are either not sensitive enough or expose the patient to ionizing radiation.

The investigators believe that hyperpolarized 129Xe MRI (HP Xe-MRI), new imaging modality, will be more sensitive then current tests and also avoid the need for ionizing radiation. To evaluate this, The investigators will compare HP Xe-MRI to PFT, when the patient is well and during a pulmonary exacerbation that is being treated.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of PCD as having either (i) biallelic mutations in known PCD genes or (ii) classic transmission electron microscopy structural ciliary defect
* Informed consent and verbal assent (as appropriate) provided by the participant's parent or legal guardian and the participant
* Ages 6-18 years and able to perform reproducible spirometry and achieve a breath hold duration sufficient for MRI acquisition

Exclusion Criteria

* Any other cardiac or respiratory disease
* Inability to perform a breath-hold of adequate duration for MRI acquisition
* Medical instability that would preclude the ability to undergo the required investigations
* FEV1 % predicted <40% on any PFT within last 2 months at time of consent
* Use of supplementary oxygen
* Severe claustrophobia
* Pregnancy or lactation
* Presence of metal implants or other MRI contraindications

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 6-18 with primary ciliary dyskinesia
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Ventilation Defect Percentage (VDP) | Within 1 year of study initiation
  Reliability; initial test
Ventilation Defect Percentage (VDP) | Within 1 week of initial test
  Reliability; re-test
Ventilation Defect Percentage (VDP) | Within 48 hours of pulmonary exacerbation diagnosis
  VDP within 48h of pulmonary exacerbation diagnosis
Ventilation Defect Percentage (VDP) | Within 48 hours of antibiotic completion
  VDP within 48h of antibiotic completion

SECONDARY OUTCOMES:
Pulmonary function tests (PFTs) | Within 1 year of study initiation
  Reliability; initial test
Pulmonary function tests (PFTs) | Within 1 week of initial test
  Reliability; re-test
Pulmonary function tests (PFTs) | Within 48 hours of pulmonary exacerbation diagnosis
  PFT within 48h of pulmonary exaction diagnosis
Pulmonary function tests (PFTs) | Within 48 hours of antibiotic completion
  PFT within 48h of antibiotic completion

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, PhD, FRCP(C), FERS, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared between two participating sites for this study. A data transfer agreement will be created and implemented to ensure smooth transfer of data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after enrolling the first participant and will be available for the duration of the study.